CLINICAL TRIAL: NCT01375530
Title: VRC 500: Screening Volunteers for Clinical Trials of Investigational Products and Licensed Products Evaluated for Research Purposes
Brief Title: Screening Volunteers for Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110164; 11-I-0164
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2025-12-19

CONDITIONS: Screening
Keywords: Prevention; Vaccine; Immunity; Evaluate; Screen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy adults 18 - 60 years old

SUMMARY:
Background:

- The National Institute of Allergy and Infectious Diseases (NIAID) at the National Institutes of Health needs healthy volunteers for vaccine clinical trials. This is a screening study that is used to identify healthy volunteers who may be eligible to participate in other clinical trials at the Vaccine Research Center that evaluate investigational vaccines, monoclonal antibodies, and injection devices. The VRC conducts studies that will allow researchers to better understand the immune system and how vaccines and monoclonal antibodies work.

Objectives:

- To screen healthy volunteers for clinical trials at the NIAID VRC.

Eligibility:

- Healthy people between 18 and 60 years of age. They must be available to take part in clinical trials and be able to provide blood for research studies.

Design:

* Screening for healthy volunteers to participate in clinical trials is an ongoing process.
* Volunteers will be asked about their medical history, including sexual activity and drug use, and a detailed physical exam will be performed.
* Blood and urine samples may be collected, and possibly other tests as needed to evaluate the volunteer's health status.
* Volunteers will not receive any investigational product in this screening protocol.

DETAILED DESCRIPTION:
The purpose of this study is to recruit and screen potential study subjects, mostly healthy volunteers, to determine if they are eligible for clinical trials of investigational products. This screening study also aims to characterize and analyze demographic information as well as laboratory and other medical findings in terms of how they may affect the eligibility of subjects for specific early phase clinical trials. All work will be conducted by the VRC Clinic of the National Institutes of Health or other IRB-approved sites that are collaborating with NIAID/VRC. Educational and recruitment materials on the investigational products and protocols will be

reviewed with and provided to subjects during participation in the screening protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: 18 years of age or older

Able and willing to complete the informed consent process

Agree to have blood and/or tissue samples collected and stored for future studies of investigational products, the immune system, and/or other medical conditions

EXCLUSION CRITERIA:

A condition in which repeated blood draws or injections pose more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access

A condition that requires active medical intervention or monitoring to avert serious danger to the participant s health or well-being

Known to be pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-08-16 (Actual)

PRIMARY OUTCOMES:
To screen subjects for their eligibility to participate in clinical trials. | Ongoing
  Duration of subject participation is variable, and may last from a few weeks to several months for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Lasonji A Holman, C.R.N.P., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Univ of MD School of Medicine Center for Vaccine Development & Global Health, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Pennsylvania-UPenn, Philadelphia, Pennsylvania

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-I-0164.html